CLINICAL TRIAL: NCT04597905
Title: Observational Study to Define Patient Preferences Toward the Attributes of Treatment Used for Inflammatory Bowel Disease, Including Efficacy Profile, Safety Profile, Frequency and Route of Administration, in Europe
Brief Title: Paricipant Preferences in the Treatment of Inflammatory Bowel Disease (IBD) in Europe
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5013; U1111-1259-3241 (Registry Identifier: WHO)
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD Participants: Participants diagnosed with CD from the 7 participating countries will take part in survey to collect data regarding their preferences towards the attributes of treatments based on DCE survey with advanced therapies for IBD, including safety and efficacy profiles, frequency and RoA in a real-world setting and data collection will be conducted in a real-world setting via an online self-reported questionnaire hosted on the Carenity platform, an international patient community.
- UC Participants: Participants diagnosed with UC from the 7 participating countries will take part in survey to collect data regarding theirpreferences towards the attributes of treatments based on DCE survey with advanced therapies for IBD, including safety and efficacy profiles, frequency and RoA in a real-world setting and data collection will be conducted in a real-world setting via an online self-reported questionnaire hosted on the Carenity platform, an international patient community.

SUMMARY:
The purpose of this survey is to describe Crohn's disease (CD) participants' as well as ulcerative colitis (UC) participants' preferences towards the attributes of treatment with advanced therapies for IBD, including safety and efficacy profiles, frequency and route of administration (RoA) in a real-world setting.

DETAILED DESCRIPTION:
This is a descriptive, observational, cross-sectional survey of participants with IBD. The survey will look into the preferences of participants towards the attributes of treatment with advanced therapies for IBD based on DCE (experimentally designed survey), including safety and efficacy profiles, frequency and RoA in a real-world setting, in European participants living with CD or UC.

The survey will involve data collection in a real-world setting via an online self-reported questionnaire hosted on the Carenity platform, an international participant community.

The survey will enroll approximately 600 participants. Participants will be enrolled in two observational cohorts:

* CD Participants
* UC Participants

This multi-center trial will be conducted in France, the United Kingdom, Italy, Spain, Belgium, Switzerland, the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported suffering from CD or UC.

Exclusion Criteria:

1. Have never been ever treated with prescription medications for CD or UC.

* Should be included in the study only once.
* Data collected from participants who subsequently withdraw their consent will not be included in or will be deleted from the database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants living with CD or UC, currently or previously treated for their condition.
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Partworth Utilities for Participants With CD and UC | 20 minutes after one time-survey start
  Partworth utilities (attribute importance scores and level values) will be evaluated separately for UC and CD in discrete choice experiment's (DCE) conditional logit (CL) models.DCEs:an attribute-based measure of benefit. CL model analyses DCEs.All DCE attributes will be included in CL models.For CD:remission after one year,occurrence of serious adverse effects or events,mild adverse effects or events, long-term remission on maintenance treatment and administration of medication.For UC: corticosteroid-free remission,healing of intestinal mucosa of bowel after one year,long-term remission on continuous treatment and administration of medication.All attributes will be coded as categorical variables;attribute levels will be dummy-coded,whereby omitted categories will be coded:0,omitted category for each attribute will be reference level of partworth utility.Negative partworth utility indicates less desired levels and positive partworth utility indicates more desired levels of attributes.

SECONDARY OUTCOMES:
Partworth Utilities for Subgroup Participants With CD and UC | 20 minutes after one time-survey start
  Partworth utilities for each pathology, by computing CL models on subgroup of participants based on demographic and medical profiles as well as quality of life criteria. Those subgroups will be created by using the clustering method available within the CL model, which will be conducted for each separated group and then compared using their estimated coefficients.
Number of Participants Categorized by Characteristics Based on Interaction With the Administration Attribute | 20 minutes after one time-survey start
Assessment of Latent Classes and Respective Partworth Utilities | 20 minutes after one time-survey start
  Latent classes and respective partworth utilities will be assessed by latent-class multinomial logit (LC-MNL) models. LC-MNL models will identify groups with similar preferences (latent classes), and estimate the probability that each respondent belongs to each class. Logistic regression models will then be applied to determine the association between latent class membership and participant characteristics.
Percentage of CD and UC Participants who Switched Their Treatment | 20 minutes after one time-survey start
Percentage of CD and UC Participants who Switched Their Treatment due to Pain | 20 minutes after one time-survey start
Mean Evaluation of Preference Rating for Intravenous Infusion | 20 minutes after one time-survey start
  Rating for intravenous infusion will be evaluated from 0 to 100 range which signifies least to most preferred.
Mean Evaluation of Preference Rating for Subcutaneous (SC) Injection With Needle and Without Needle | 20 minutes after one time-survey start
  Rating for SC injection will be evaluated from 0 to 100 range which signifies least to most preferred.
Mean Evaluation of Preference Rating For Oral Tablet or Pill | 20 minutes after one time-survey start
  Rating for tablet/pills will be evaluated from 0 to 100 range which signifies least to most preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Carenity, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/